CLINICAL TRIAL: NCT01199406
Title: Combined Preincisional Infiltration and Intraperitoneal Instillation of Levobupivacaine for Postoperative Pain Reduction After Laparoscopic Cholecystectomy; A Double-blind Placebo-controlled Randomised Clinical Trial
Brief Title: Pain Reduction After Cholecystectomy
Acronym: INTENSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meander Medical Center (Other)
Responsible Party: dr. Consten, Meander medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Intense Trial
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Cholecystolithiasis; Postoperative Pain
Keywords: gallstone; gallbladder; cholecystectomy; laparoscopic; pain
MeSH Terms: conditions — Cholecystolithiasis; Pain, Postoperative; Gallstones; Pain | interventions — Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- normal saline (Placebo Comparator): 80 mL 0.9% NaCl
  Interventions: Drug: Levobupivacaine
- Levobupivacaine (Experimental): 80mL 0.125% levobupivacaine
  Interventions: Drug: Levobupivacaine

INTERVENTIONS:
Drug: Levobupivacaine — 0.125% levobupivacaine 80 mL (100 mg) intraoperative, 20 mL subcutaneously and 60 mL intraperitoneally
  Other Names: Chirocaine (brand name); NDA 20-997

SUMMARY:
To determine the effect of combined intracutaneous infiltration and intraperitoneal instillation of 80 mL 0,125% levobupivacaine prior to the start of laparoscopic cholecystectomy on abdominal pain up to 24 hours after surgery.

DETAILED DESCRIPTION:
The primary endpoint of this study was postoperative abdominal pain as measured by a visual analogue scale (VAS), using a VAS lineal with a slide. The patient was asked to indicate a score from 0 to 100 corresponding to his or her pain. At 0.5, 2, 4, 8 and 24 hours after the surgical procedure the primary investigator visited the patient to obtain the VAS scores.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 80
* ASA I or II
* with symptomatic gallstone disease which requires elective laparoscopic cholecystectomy

Exclusion Criteria:

* acute cholecystitis, cholangitis, severe acute pancreatitis, advanced liver cirrhosis or suspected gallbladder cancer,
* a medical history of epilepsy, cardiac arrhythmias or chronic pain of any kind, - allergy to amid type drugs
* pregnancy
* patients suffering from hypotension or hypovolemia
* infectious liver disease
* conditions obstructing adequate pain scoring
* patients using drugs that deduce function of the CYP3A4 or CYP1A2 system
* patients having an American Society of Anaesthesiologists (ASA) classification of three or higher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Abdominal Pain in Visual Analogue Scale (VAS 0-100mm) | 24 h postoperatively
  Postoperative abdominal pain

SECONDARY OUTCOMES:
Shoulder pain | 24 h
  Postoperative shoulder pain
Rescue Analgesics | 24 h postoperatively
  The need of rescue analgesics within the 24h postoperatively
adverse events caused by the investigational procedure or by levobupivacaine itself | Intra- and postoperative up to 24 hours
  Adverse events were defined as neurological or cardial effects attributable to use of levobupivacaine. Adverse events by the procedure such as bleeding were also registered.
Length of hospital stay | Maximum two weeks
intra-operative complications including perforation of the gallbladder, bile duct injury, bowel injury and injury to vascular structures | intraoperative, 1 hour
postoperative complications during hospitalisation | during hospitalisation (up to two weeks)
  Infection, bleeding, embolisation etc.

CONTACTS AND LOCATIONS:
Overall Officials: Werner A Draaisma, MD, PhD, Study Chair — Meander MC; Bart Hilvering, MD, Principal Investigator — Meander MC; Esther CJ Consten, MD, PhD, Study Director — Meander MC; Kristine E Kofman, MD, Study Chair — Meander MC; Rene M Valk, MD, Study Chair — Meander MC; Jarmila DW Van der Bilt, MD, Study Chair — Meander MC
Locations (1):
- Meander MC, Amersfoort, Amersfoort, Netherlands

REFERENCES:
- [Derived] Hilvering B, Draaisma WA, van der Bilt JD, Valk RM, Kofman KE, Consten EC. Randomized clinical trial of combined preincisional infiltration and intraperitoneal instillation of levobupivacaine for postoperative pain after laparoscopic cholecystectomy. Br J Surg. 2011 Jun;98(6):784-9. doi: 10.1002/bjs.7435. Epub 2011 Mar 17. PMID 21412996